CLINICAL TRIAL: NCT04725734
Title: Air Pollution and Daily Mobility of Pregnant Women in the Eurometropole: Identification of Critical Windows of Exposure During Pregnancy
Brief Title: Air Pollution and Daily Mobility of Pregnant Women Identification of Critical Windows of Exposure
Acronym: MOBIFEM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8000
Record Dates: First submitted 2020-10-05; First posted 2021-01-27 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Pregnancy; Low Birth Weight; Preterm Birth; Air Pollution
Keywords: social inequalities
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Pregnant women — The patients will complete a questionnaire for each quarter

SUMMARY:
This study is conducted to assess the role of pregnant women's daily mobility living in the Eurometropole of Strasbourg in a context of the existence of environmental exposure disparities (PM10, PM2.5, NO2). Furthermore, this study will tend to identify the critical windows of exposure and of greater risk of the adverse pregnancy outcomes as low birth weight and prematurity.

A second question addressed in this work is to assess the relationship between the pregnant women's socio-economic status and the air pollution exposure (PM10, PM2.5, NO2).taking into account the spatio-temporal variations of the exposure as well as the critical windows of exposure during pregnancy.

The present work deals with the following question "how does the combination of environmental exposure, socio-economic status and women's daily mobility, could contribute to socio-spatial inequalities in the health of the newborn? The underlying hypothesis is that the accumulation, in given area, of environmental exposures (as PM10, PM2.5 and NO2), of unfavorable living conditions (socio-economic environment) and individual factors (specific spatio-temporal trajectory) would induce an increased risk for the health of the newborn, (more particularly in terms of birth weight and term of birth). This hypothesis is structured 4 sub-hypotheses: i) The misclassification of exposure is socially distributed among pregnant women living in the Eurometropole of Strasbourg. ii) Beyond maternal and fetal characteristics, pregnant women who reside in a more socio-economically deprived neighborhood and / or with higher levels of environmental exposure to PM10, PM2.5 and NO2 are more at risk of preterm newborn and low birth weight newborn. iii) The accumulation of environmental exposures of the pregnant women and their daily mobility over their territory during the pregnancy increase the health inequalities of the newborn. iv) The critical windows of fetal exposure to pollutants is related to the socioeconomic level of their neighborhood and to the daily mobility of the women in their territory during pregnancy. Women are included in the study at the time of their first or second trimester ultrasound. Here are the tools used in the study: Descriptive survey of their idividuals characteristics, descriptive survey of women's mobility to assess their exposure during each trimester of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women dwelling in the Eurometropole of Strasbourg
* Women who have done ultrasound monitoring in the HUS (Hopitaux Universitaires de Strasbourg)
* Good understanding of the French language
* Women who give her signed agreement of non-opposition to research and / or who give her signed consent for the data collect

Non-inclusion criteria:

* refusal to participate in the study
* under-age women (<18 years old)
* women who not have a clear understanding of the information (emergency situation, comprehension problems…)
* Women must not be under tutorship or curatorship or under the protection of a conservator ("sauvegarde de justice")

Exclusion criteria:

* premature delivery threats
* placenta previa
* twin pregnancy
* pre-eclampsia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women, include at 1st or 2nd trimester in the Hautepierre and CMCO ultrasound department.
  The period of inclusion should extend from 1 October 2020 to 31 October 2021 with a duration of participation of each subject of 9 months.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-02-04 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Characteristics of the newborn | 7 months
  Estimation of fetal weight
Characteristics of the newborn | 7 months
  Estimation of birth weight

CONTACTS AND LOCATIONS:
Overall Officials: Virginie HAMANN, Principal Investigator — Les Hôpitaux Universitaires
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Schiltigheim, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Simoncic V, Hamann V, Huber L, Deruelle P, Sananes N, Enaux C, Alter M, Schillinger C, Deguen S, Kihal-Talantikite W. Study protocol to explore the social effects of environmental exposure and lifestyle behaviours on pregnancy outcome: an overview of cohort of pregnant women study. BMJ Open. 2022 Sep 17;12(9):e058883. doi: 10.1136/bmjopen-2021-058883. PMID 36115665